CLINICAL TRIAL: NCT03290144
Title: Occurrence of Pregnancies in Women With Cystic Fibrosis
Brief Title: Pregnancies and Cystic Fibrosis
Acronym: MUCOG
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0624
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis - Pregnancy - Diabetes
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with diabetes
- without diabetes

SUMMARY:
There have been substantial advances in care for individuals with CF, including improved nutrition and respiratory care. Women with CF are now likely to survive into adulthood with a median predicted survival of 49.7 years in 2012, which have resulted in increasingly normal lifestyles, including successful pregnancies in women with CF. The number of pregnancies in CF women has increased as reported by the 2013 Annual Data Report from the French CF Registry (6 pregnancies in 1992 to 53 in 2012). Pregnancy adds many physiological stresses to the body, particularly on pulmonary function (decrease in residual volume, expiratory reserve capacity) and nutritional status (increase in nutritional needs). In women with CF, these added stresses could theoretically affect survival, with difficulties to maintain adequate nutrition and an unpredictable effect on lung function. A number of studies published over the past 15 years have attempted to clarify the risk of pregnancy in women with CF to guide clinicians and women. Many authors compared the outcomes of pregnant CF women to non-pregnant CF women regardless of nutritional status, lung function, diabetes mellitus, bacteriological colonization. In literature, pregnancy was possible and well tolerated in CF women with mild disease if associated with more intensive monitoring and aggressive treatment during pregnancy, with particular emphasis on nutrition and weight gain. CF women have an increased likelihood of receiving treatment for diabetes both during and after pregnancy. Furthermore diabetes mellitus has been associated with more severe pulmonary disease, more frequent pulmonary exacerbations, poorer nutritional status and a reduced life expectancy. Pre-pregnancy diabetes mellitus is associated with a poorer prognosis for pregnancy in general population. Severe forms of CF, including pre-pregnancy diabetes mellitus might as well do badly with accelerated decline after pregnancy. To determine the effect of pre-pregnancy diabetes on maternal decline after pregnancy, we will compare FEV1 and BMI rates of decline, during a two-years follow-up period after pregnancies, reported in the French CF Registry, according to their diabetic status.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis women attending the CF French Registry between January 1, 2001 and December 31, 2010

Exclusion Criteria:

* Women who had received a pulmonary graft before pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pregnant, Cystic Fibrosis (CF) women attending the CF French Registry between January 1, 2001 and December 31, 2010.
Enrollment: 450 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2018-09-02 (Estimated); Study Completion 2018-09-02 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 | 12 months following the pregnancy

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | 12 months following the pregnancy

IPD SHARING:
Plan to Share IPD: No